CLINICAL TRIAL: NCT01150136
Title: Choline Nutritional Status Of Children With Cystic Fibrosis X-Sectional Study
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: H07-01140
Record Dates: First submitted 2010-04-26; First posted 2010-06-24 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Cystic Fibrosis
Keywords: choline; cystic fibrosis; methyl metabolism; oxidative stress
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children with proven CF and known genotype, age 0-17 yr

SUMMARY:
Cystic fibrosis (CF) is the most common lethal, inherited disorder among Caucasians. Choline is an essential vitamin and as a methyl donor is critically needed to support the normal metabolism. Our previous studies have demonstrated that children with CF have depleted levels of choline. The purpose of this study is to gather data on the status of choline and related metabolites in children with Cystic Fibrosis by age and gender. The hypothesis for this study is that in children with CF, deficiency of choline and related metabolites will increase with increasing age.

DETAILED DESCRIPTION:
The objective of this clinical project is to determine the status of choline and related metabolites in a large group of children with Cystic Fibrosis (CF). Based on the results it will be possible to determine which children are deficient or at risk for choline deficiency, and might benefit most from supplementation to sustain improvement in the plasma choline, and its metabolites. This will be a cross-sectional study that will, over a 6 month period, look to enroll as many patients as possible from 140 children with CF who are seen regularly at the CF Clinic at B.C.'s Children's Hospital. The study will involve the collection of blood and urine at the time of a scheduled appointment. All procedures for enrollment, collection of chart data and blood samples will follow procedures used in our previous studies. Body weight and height will be measured and routine blood work including liver enzymes, hematology, serum zinc, selenium and vitamins A and E will be completed as part of the clinic appointment. CF genotype, gender, birth date, hematology, clinical chemistry, anthropometric and nutritional measures, liver ultrasound, biopsy reports where available, pancreatic function (elastase, chymotrypsin/secretin-CCK) and all medications including mineral, vitamin and nutritional and enzyme supplements will be recorded from chart data. Blood samples will be used for analyses of choline and its metabolites and various biomarkers in redox pathways. A urine sample will be collected and used to assay excretion of related metabolites. Creatine will be analyzed to avoid the need for quantitative 24 hour urine collection.

ELIGIBILITY:
Inclusion Criteria:

* children with proven CF and known genotype.
* age 0-17 yr.
* outpatients of the CF Clinic at the British Columbia (B.C.) Children's Hospital.
* Children without CF or any other known disease.

Exclusion Criteria:

* children with CF receiving parenteral nutrition during the previous week.
* children who are hospitalized.
* children with any health problems other than CF that might in the opinion of the investigators influence dietary choices, growth, choline or methyl metabolites.

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with proven CF and known genotype, age 0-17 yr who are outpatients of the CF Clinic at the British Columbia (B.C.) Children's Hospital
Sampling Method: Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2007-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
The change in plasma choline and its metabolites with increasing age in children with CF compared to a healthy reference group without CF | 12 months

SECONDARY OUTCOMES:
The relationship between choline and acetylcholine, and markers of oxidative stress, inflammation and disturbed methyl metabolism | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M. Innis, Dr., Principal Investigator — University of British Columbia; A. George F. Davidson, MD, Study Director — University of British Columbia
Locations (1):
- Child & Family Research Institute, CF Clinic, BC Children's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Innis SM, Davidson AG, Bay BN, Slack PJ, Hasman D. Plasma choline depletion is associated with decreased peripheral blood leukocyte acetylcholine in children with cystic fibrosis. Am J Clin Nutr. 2011 Mar;93(3):564-8. doi: 10.3945/ajcn.110.005413. Epub 2011 Jan 12. PMID 21228267